CLINICAL TRIAL: NCT07029893
Title: Independent Life Skills Program for Adults With Autism Spectrum Disorder: A Pilot Randomized Controlled Trial
Brief Title: Independent Life Skills Program for Adults With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LIU Karen, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HongKongPU_IndependentLifeSkil
Record Dates: First submitted 2025-06-10; First posted 2025-06-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; Independent living skills; Pilot randomized controlled trial
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Independent Life Skills Program (ILSP) (Experimental): 14-week Independent Life Skills Program (ILSP)
  Interventions: Behavioral: Independent Life Skills Program (ILSP)
- Wait-list control (Sham Comparator): Wait-list control - participants do not receive intervention
  Interventions: Other: Wait-list control

INTERVENTIONS:
Behavioral: Independent Life Skills Program (ILSP) — The ILSP runs for 14 weeks, covering six areas of independent living skills and 14 weekly sessions lasting 2 hours each. The program will run in a group format with 4 participants in each group. The ILSP will be run by occupational therapists who are trained in the program delivery.
  Arms: Independent Life Skills Program (ILSP)
Other: Wait-list control — Participants do not receive the experimental treatment and will be put on a waiting list to receive the intervention after the active treatment group does.
  Arms: Wait-list control

SUMMARY:
This project will pilot-test an Independent Life Skills Program (ILSP) for people with Autism Spectrum Disorder. The ILSP was developed by a group of occupational therapists at Heep Hong Society based on the theories of self-regulated learning, life management, and self-management. The ILSP is a comprehensive program covering different life skills, including personal management, home management, community integration and self-management. These life skills are essential for transitioning from young adulthood and are predictors of successful transition.

DETAILED DESCRIPTION:
Acquiring daily life skills, including personal management, home management, community integration, and self-management, is crucial for enhancing quality of life and promoting autonomous living. However, individuals with Autism Spectrum Disorder (ASD), encompassing both adolescents and adults, often face challenges and demonstrate limited levels of independence when it comes to engaging in these daily living skills.

This pilot testing aims to investigate the feasibility and acceptability of the ILSP for individuals with ASD. It will also pilot-test the benefits of daily living skills and confidence.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or above;
* diagnosed with autism based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* borderline to normal IQ.

Exclusion Criteria:

* have other types of Special Educational Needs such as social and emotional mental health needs, hearing impairments
* do not consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Goal Attainment Scaling (GAS) | Before the intervention period, and at the end of the intervention period at 14 weeks
  The GAS takes into account that individuals have varying starting points and different desired outcomes based on their unique strengths and challenges. It is proven to be useful in reflecting personalised outcomes in intervention studies for adults with autism. The GAS uses a 5-point scale to create goals and measure progress, with -2 representing the baseline skill level. Progression from -2 to -1 indicates progress (50% better performance), and progression from -2 to 0 indicates the expected level of outcome (100% better performance).

SECONDARY OUTCOMES:
Instrumental Activities of Daily Living (IADL) Confidence Questionnaire | Before the intervention period, and at the end of the intervention period at 14 weeks
  This questionnaire was designed by the occupational therapists. It covers the six areas of the ILSP. Participants will be asked to rate their confidence in completing those six areas and 14 skills using an 11-point scale, from 0 as no confidence at all to 10 as full confidence. The minimum score is 0 and the maximum score is 300.
IADL Competency Test | Before the intervention period, and at the end of the intervention period at 14 weeks
  Based on the content of the ILSP, the occupational therapists developed this competency test to assess participants' competence in 30 skills. The minimum score is 0 and the maximum score is 30.
Lawton Instrumental Activities of Daily Living Scale - Hong Kong version (IADL Scale) | Before the intervention period, and at the end of the intervention period at 14 weeks
  It covers nine complex daily tasks (IADL) needed to live independently (e.g., doing housework, preparing meals, taking medications properly, managing finances, using a telephone). A 4-point scoring system is used with 0, representing unable to perform to 3 representing complete independence. The score ranges from 0 - 27, with lower scores indicating less ability to complete the daily tasks.

OTHER OUTCOMES:
Acceptability survey | At the end of the intervention at 14 weeks
  The survey will be completed by participants in the ILSP (experimental intervention). Questions in the survey are based on four dimensions to determine the participants' preparedness to participate, relevancy, convenience and perceived effectiveness of the ILSP. The questionnaire uses a four-point Likert scale with verbal labels indicating equal graduating portions of agreement or disagreement from (1) completely disagree, (2) disagree, (3) agree, and (4) completely agree.
Attendence rate | Through intervention completion, attendence of every session in the 14-week intervention
  Participants' retention rate and attendance in each session are recorded and a percentage attendance rate is calculated to reflect the program's feasibility. This is recorded for participants in the ILSP (experimental intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Liu, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The project is considering applying for external funding. The IPD may be shared after the funding application announcement and after data collection.